CLINICAL TRIAL: NCT00189748
Title: An Extension Study of the Patients Enrolled in Acute Graft Versus Host Disease (GVHD) Prophylaxis Study (Protocol No. FJ-506E-BT01) to Assess Safety and Efficacy of GVHD Prophylaxis of a Tacrolimus New Oral Formulation (MR4).
Brief Title: A Study to Assess the Safety and Efficacy of a Tacrolimus New Oral Formulation (MR4) in BMT Patients-Extension-
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ-506E-BT02
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Bone Marrow Transplantation; Graft Versus Host Disease; Graft-Versus-Host Disease; Graft-Vs-Host Disease
Keywords: Tacrolimus; Immunosuppression; Bone Marrow Transplantation; Graft versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus

SUMMARY:
To assess safety and efficacy of the patients with MR4 therapy in GVHD prophylaxis study who are eligible for the administration after 100 days post transplant (up to 1 year)

ELIGIBILITY:
Inclusion Criteria:

* Patient had enrolled in GVHD prophylaxis study.
* Patient had been fully informed.

Exclusion Criteria:

* The patient had been not eligible for the administration after 100 days post transplant in the investigator's judgement.

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Clinical development, Study Chair — Astellas Pharma Inc., Japan
Locations (4):
- Japan (4):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kyusyu Region